CLINICAL TRIAL: NCT00483145
Title: Laser-Mediated Photodynamic Therapy of Acne Vulgaris and Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Merete Hædersdal, Bispebjerg Hospital
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: KF-01-328309
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Acne Vulgaris and Rosacea
MeSH Terms: conditions — Acne Vulgaris; Rosacea

ARMS (2):
- 1 (Active Comparator): Long-pulsed dye laser (Candela)
  Interventions: Device: Long-pulsed dye laser (Candela) and PDT (methylaminolevulinate); Device: Long-pulsed dye laser
- 2 (Active Comparator): Long-pulsed dye laser assisted fotodynamic therapy (methylaminolevulinate)
  Interventions: Device: Long-pulsed dye laser (Candela) and PDT (methylaminolevulinate); Device: Long-pulsed dye laser assisted fotodynamic therapy (methylaminolevulinate)

INTERVENTIONS:
Device: Long-pulsed dye laser (Candela) and PDT (methylaminolevulinate)
Device: Long-pulsed dye laser
  Arms: 1
Device: Long-pulsed dye laser assisted fotodynamic therapy (methylaminolevulinate)
  Arms: 2

SUMMARY:
To evaluate efficacy and adverse effect from long-pulsed dye laser versus long-pulsed dye laser-mediated photodynamic therapy for acne vulgaris and rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory acne and rosacea
* Skin types I-IV

Exclusion Criteria:

* Patients younger than 18 years
* Skin types V and VI
* Topical and systemic conventional acne treatments

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark